CLINICAL TRIAL: NCT03701464
Title: Comparison of Clinical Efficacy Between ENGBD and PTGBD in Acute Suppurative Cholecystitis: a Single-center, Prospective Randomized Trial
Brief Title: Comparison of ENGBD and PTGBD in Acute Suppurative Cholecystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENGBD in acute cholecystitis
Record Dates: First submitted 2018-10-05; First posted 2018-10-10 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Success Rate
Keywords: ERCP; PTGBD; ENGBD; Gallbladder drainage; Cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic naso-gallbladder drainage (Experimental): After selective bile duct cannulation, a 0.025- or 0.035-inch guidewire is advanced into the cystic duct and subsequently into the gallbladder. A 5F naso- Pancreas catheter was inserted into the gallbladder for ENGBD.
  Interventions: Procedure: Endoscopic naso-gallbladder drainage
- Percutaneous gallbladder drainage (Active Comparator): Ultrasound guided，an 18-gauge needle is inserted into the gallbladder，0.035 inch guidewire is coiled into the gallbladder and 9Fr dilator expands the skin,then 8Fr-20cm catheter is placed.
  Interventions: Procedure: Percutaneous gallbladder drainage

INTERVENTIONS:
Procedure: Endoscopic naso-gallbladder drainage — Using ERCP technique insert a naso-gallbladder drainage tube through common bile duct and cystic duct.
  Arms: Endoscopic naso-gallbladder drainage
Procedure: Percutaneous gallbladder drainage — Percutaneous transhepatic technique insert drainage tube into gallbladder
  Arms: Percutaneous gallbladder drainage

SUMMARY:
Comparison of ENGBD and PTGBD methods on clinical outcomes and the difficulty of cholecystectomy in later stage in patients with acute suppurative cholecystitis.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy was the standard surgical method for acute cholecystitis unless difficulty in resection due to acute inflammation, no improvement after supportive therapy, or early inability to tolerate cholecystectomy. In this setting, gallbladder drainage was needed. Percutaneous transhepatic gallbladder drainage (PTGBD)was used as a first-line mitigation method, whose restrictions are contraindications and strong pain caused by puncture. Endoscopic technique based on endoscopic retrograde cholangiopancreatography (ERCP) had been made another alternative management for drainage. Endoscopic drainage expanded the indications for drainage without reducing the technical success rate and clinical remission rate, especially less uncomfortable, which greatly improved the quality of life for patients. Unfortunately, because of the difficult procedures and long learning curve, endoscopic gallbladder drainage can only be performed in some large endoscopic centers. Despite a few prospective comparison of PTGBD and endoscopic ultrasound EUS drainage studies so far, there is no prospective study comparing endoscopic naso-gallbladder drainage （ENGBD） and PTGBD, especially in its impacts while cholecystectomy. This study aim to observe clinical effects of ENGBD and PTGBD during the all stage of peri-cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Acute suppurative cholecystitis
* Who can not tolerate or unsuitable for cholecystectomy

Exclusion Criteria:

* Unwillingness or inability to consent for the study
* Coagulation dysfunction (INR> 1.5) and low peripheral blood platelet count (<50×10^9 / L) or using anti-coagulation drugs
* Bile duct stones
* Prior surgery of Bismuth Ⅱ, Roux-en-Y and Cholangiojejunostomy
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage or perforation, severe liver disease(such as decompensated liver cirrhosis, liver failure and so on), septic shock
* Any malignant
* Pregnant women or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Pain remission（visual-analogue scale） | 3 weeks
  Pain assessment would be performed using the visual-analogue scale after procedures. Draw a 10 cm line on a piece of paper, mark one end of the line with the nubmer 0, indicating no pain; the other end with 10, indicating severe pain; the middle part indicates different degrees of pain. While assesing the pain scale, make sure the patient can not see the numbers on the paper, and let them mark the position according to their feelings about the pain. And the physician will have a score based on the mark.

SECONDARY OUTCOMES:
Gallbladder drainage success rate | 3 months
  Bile juice outflow more than 50ml a day
Migration | 3 months
  Number of participants with tube dislocation from gallbladder
Hemorrhage | 3 months
  Number of participants with bleeding which was defined as hemoglobin deceased, or required transfusion or additional intervention
Perforation | 3 months
  Number of participants whose CT scan shows retroperitoneal or gallbladder space fluid or gas
Bile leak | 3 months
  Number of participants with bile juice leak into abdomen
Number of participants with Pancreatitis | 3 months
  Was defined as typical pain, Serum amylase at least three times than normal after EPCP
Cholecystectomy duration | 3 months
  Time of laparoscopic cholecystectomy
Hemorrhage during cholecystectomy | 3 months
  The amount of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, MD,PhD, Study Director — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jang JW, Lee SS, Song TJ, Hyun YS, Park DY, Seo DW, Lee SK, Kim MH, Yun SC. Endoscopic ultrasound-guided transmural and percutaneous transhepatic gallbladder drainage are comparable for acute cholecystitis. Gastroenterology. 2012 Apr;142(4):805-11. doi: 10.1053/j.gastro.2011.12.051. Epub 2012 Jan 11. PMID 22245666
- [Background] Kedia P, Sharaiha RZ, Kumta NA, Widmer J, Jamal-Kabani A, Weaver K, Benvenuto A, Millman J, Barve R, Gaidhane M, Kahaleh M. Endoscopic gallbladder drainage compared with percutaneous drainage. Gastrointest Endosc. 2015 Dec;82(6):1031-6. doi: 10.1016/j.gie.2015.03.1912. Epub 2015 May 5. PMID 25952093
- [Background] Itoi T, Kawakami H, Katanuma A, Irisawa A, Sofuni A, Itokawa F, Tsuchiya T, Tanaka R, Umeda J, Ryozawa S, Doi S, Sakamoto N, Yasuda I. Endoscopic nasogallbladder tube or stent placement in acute cholecystitis: a preliminary prospective randomized trial in Japan (with videos). Gastrointest Endosc. 2015 Jan;81(1):111-8. doi: 10.1016/j.gie.2014.09.046. PMID 25527052
- [Background] Khan MA, Atiq O, Kubiliun N, Ali B, Kamal F, Nollan R, Ismail MK, Tombazzi C, Kahaleh M, Baron TH. Efficacy and safety of endoscopic gallbladder drainage in acute cholecystitis: Is it better than percutaneous gallbladder drainage? Gastrointest Endosc. 2017 Jan;85(1):76-87.e3. doi: 10.1016/j.gie.2016.06.032. Epub 2016 Jun 22. PMID 27343412
- [Derived] Mu P, Lin Y, Zhang X, Lu Y, Yang M, Da Z, Gao L, Mi N, Li T, Liu Y, Wang H, Wang F, Leung JW, Yue P, Meng W, Zhou W, Li X. The evaluation of ENGBD versus PTGBD in high-risk acute cholecystitis: A single-center prospective randomized controlled trial. EClinicalMedicine. 2020 Dec 23;31:100668. doi: 10.1016/j.eclinm.2020.100668. eCollection 2021 Jan. PMID 33385126
- [Derived] Mu P, Yue P, Li T, Bai B, Lin Y, Zhang J, Wang H, Liu Y, Yao J, Meng W, Li X. Comparison of endoscopic naso-gallbladder drainage and percutaneous transhepatic gallbladder drainage in acute suppurative cholecystitis: Study Protocol Clinical Trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Feb;99(8):e19116. doi: 10.1097/MD.0000000000019116. PMID 32080085